CLINICAL TRIAL: NCT06541873
Title: DuALS - A Cross-sectional Observational Study of Gait Patterns in Dual-task Conditions in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Gait Patterns in Dual-task Conditions in Patients With Amyotrophic Lateral Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, MD, Professor, IRCCS San Raffaele
Other Study IDs: DuALS
Record Dates: First submitted 2024-07-08; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ALS or other motor neuron disease phenotype: Patients with ALS and other MND phenotypes will undergo gait evaluation using wearable sensors in different conditions (single-task vs dual-task conditions).
  Interventions: Other: Clinical and gait evaluation
- Healthy controls: 30 healthy controls with similar age and sex distribution will undergo the same evaluations as patients
  Interventions: Other: Clinical and gait evaluation

INTERVENTIONS:
Other: Clinical and gait evaluation — The dual-task conditions to be assessed during gait performance will include: counting backwards by 3 (executive simple task); counting backwards by 7 (executive complex task); mnemonic recall of the Rey's Auditory Verbal Learning Test (RAVLT). Performance scores will be correlated with cognitive status and clinical features. Data will be collected at the baseline (i.e., only) visit within the enrollment timeframe of 3 years from study initiation.

SUMMARY:
The investigators hypothesize a relevant impact of cognitive status over gait performance in patients with amyotrophic lateral sclerosis (ALS), contributing to poor mobility and representing a relevant risk for falls. The present observational, cross-sectional study on ambulatory patients with ALS will evaluate gait performance using different sets of dual-task conditions to demonstrate the importance of cognitive aspects in rehabilitation programs for these patients. The dual-task conditions to be assessed during gait performance will include: counting backwards by 3 (executive simple task); counting backwards by 7 (executive complex task); mnemonic recall of the Rey's Auditory Verbal Learning Test (RAVLT). Patients' performance will be compared with a group of healthy controls with similar age and sex distribution in order to highlight the specific effects of the disease.

ELIGIBILITY:
Patient inclusion criteria:

* Age ≥ 18 years;
* Clinical diagnosis of ALS or other MND phenotype;
* Able to walk unassisted for at least 1 minute consecutively;
* Oral and written informed consent to study participation.

Healthy control inclusion criteria:

1. Age ≥ 18 years;
2. Age and sex distribution similar to patients (age range: mean age of patients years ± 15 years);
3. Able to walk unassisted for at least 1 minute consecutively;
4. Oral and written informed consent to study participation.

Exclusion Criteria

An individual (either patient or healthy control) who meets any of the following criteria will be excluded from participation in this study:

1. Diagnosis of dementia;
2. Medical conditions or substance abuse that could interfere with cognition;
3. Any (other) major systemic, psychiatric, neurological, visual, and musculoskeletal disturbances or other causes of walking inability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Based on previous experience and referral rates to the San Raffaele ALS Center (directed by the PI, including the Neurology and Neurorehabilitation wards and outpatient ALS clinic counting 50 new patients/year, 80 second opinion/year; 120 patients in care), the investigators plan to enroll at least 30 patients with ALS or any other MND phenotype, as well as 30 healthy controls with similar age and sex distribution, in line with sample size of previous studies ranging from 11 (Hausdorff et al., 2000) to 42 (Dubbioso et al., 2023). Healthy controls will be recruited by word of mouth, via consenting friends and non-consanguineous relatives who will be accompanying patients for study visits. Subjects will be assessed for suitability from their clinical notes or via a telephone screen. Given the cross-sectional, single-visit design of the present study, the investigators expect all patients to complete the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Dual-task cost at 1-Minute Walking Test performance | Cross-sectional (baseline) evaluation
  Percentage of variability of gait scores obtained at the 1-Minute Walking Test (1minWT) (i.e., meters walked in one minute) in dual-task vs. single-task conditions in ALS patients compared with healthy controls
Dual-task cost at Timed Up and Go performance | Cross-sectional (baseline) evaluation
  Percentage of variability of gait scores obtained at the Timed Up and Go (TUG) test (i.e., time in seconds) in dual-task vs. single-task conditions in ALS patients compared with healthy controls

SECONDARY OUTCOMES:
Walking velocity | Cross-sectional (baseline) evaluation
  Performance at 10 Meters Walking Test (10MWT) in terms of time (seconds)
Executive simple task | Cross-sectional (baseline) evaluation
  Ability to count backwards by 3 (number of correct subtractions in one minute)
Executive complex task | Cross-sectional (baseline) evaluation
  Ability to count backwards by 7 (number of correct subtractions in one minute)
Mnemonic ability | Cross-sectional (baseline) evaluation
  Performance at Rey's Auditory Verbal Learning Test (RAVLT) (number of correct immediate recalls of 15 items presented verbally).
Functional disability | Cross-sectional (baseline) evaluation
  ALS Functional Rating Scale scores [ALSFRS-r] ranging from 0 (worst functional status) to 48 (best functional status), as available from clinical charts
Muscle strength | Cross-sectional (baseline) evaluation
  Medical Research Council [MRC] muscle testing in each tested muscle district ranging from 0 (worst performance) to 5 (best performance), as available from clinical charts
Cognitive impairment | Cross-sectional (baseline) evaluation
  Edinburgh Cognitive Assessment Scale [ECAS] performance ranging from 0 (worst performance) to 136 (best performance), as available from clinical charts

IPD SHARING:
Plan to Share IPD: No